CLINICAL TRIAL: NCT04932460
Title: A Prospective Multi-center Study: Contrast-enhanced Ultrasonography Combined With Blue Dye as Dual-tracer for Sentinel Lymph Node Biopsy After Neoadjuvant Therapy in Breast Cancer
Brief Title: Contrast-enhanced Ultrasonography Combined With Blue Dye as Dual-tracer for Sentinel Lymph Node Biopsy
Acronym: Asclepius
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: The Seventh Affiliated Hospital of Sun Yat-sen University (Other); Affiliated Hospital of Guangdong Medical University (Other); First Affiliated Hospital of Shantou University Medical College (Other)
Responsible Party: Principal Investigator, Ying Lin, Vice Director of Department of Breast Surgery, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021332GD
Record Dates: First submitted 2021-05-31; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Breast Neoplasms; Neoadjuvant Therapy; Sentinel Lymph Node Biopsy
Keywords: contrast enhanced ultrasonography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CEUS+blue dye (Experimental): The included patients will accept essential tests and CEUS before and after neoadjuvant chemotherapy to evaluate axillary lymph nodes status. When patients finish neoadjuvant therapy, SLNB with or without axillary lymph node dissection will be performed using CEUS lymphatic mapping to mark SLN on the skin combined with blue dye.
  Interventions: Procedure: CEUS; Procedure: blue dye

INTERVENTIONS:
Procedure: CEUS — CEUS is performed before neoadjuvant treatment and surgery to evaluate the status of axillary lymph node and locate the sentinel lymph node.
Procedure: blue dye — Before operation, blue dye is injected for sentinel lymph node mapping.

SUMMARY:
False negative rate (FNR) in patients who has accepted neoadjuvant therapy is high. Blue dye and radioisotope as dual-tracer can decrease FNR. Several large clinical trials showed that using dual trace with blue dye and radioisotope can reduce the FNR to less than 10%. But radioisotope is still not approved in China and can cause radiocontamination. A novel dual-tracer which can decrease the FNR in patients after neoadjuvant therapy is urged to be explored. Contrast enhanced ultrasonography (CEUS) can make the lymphatic drainage path and sentinel lymph nodes visible. Retrospective studies found that CEUS can locate SLN precisely. So this clinical trial aim to evaluate FNR, detective rate and numbers of SLN by using CEUS combined with blue dye as dual-tracer in sentinel lymph node biopsy in breast cancer patients after neoadjuvant therapy and the accuracy of CEUS for the diagnosis of lymph node metastasis before and after neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old female；
* ECOG：0 - 1；
* Biopsy confirmed invasive breast cancer；
* cT1-4N0-3；
* Signed informed consent.

Exclusion Criteria:

* Inflammatory breast cancer；
* Received ipsilateral axillary surgery previously；
* During pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 350 (Estimated)
Dates: Start 2021-06-15 (Estimated); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
False negative rate | 6 months
  The false negative rate (FNR) of sentinel lymph node biopsy using dual-tracer with CEUS and blue dye after neoadjuvant chemotherapy in invasive breast cancer patients.
  The FNR is calculated as the number of false negative cases divided by the number of false negative plus true positive cases and then multiplied by 100%.

SECONDARY OUTCOMES:
The detective rate of sentinel lymph node biopsy | 6 months
  The detective rate of SLNB after neoadjuvant therapy when using blue dye and CEUS lymphatic mapping as dual tracer.
  The detective rate is calculated as the number of patients in whom SLN can be detected during SLNB divided by the number of patients with the treatment of SLNB and then multiplied by 100%.
The average numbers of sentinel lymph node | 6 months
  The average numbers of sentinel lymph node is calculated as the number of all SLNs detected during SLNB divided by the number of patients received SLNB and then multiplied by 100%.
The accuracy of CEUS in evaluation of axillary lymph nodes in breast cancer | 6 months
  The accuracy of CEUS in evaluation of axillary lymph nodes in breast cancer patients before and after neoadjuvant therapy.
  The accuracy rate is calculated as the number of true positive plus true negative cases divided by the number of patients then multiplied by 100%.

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of Sun Yat-Sen university, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kuehn T, Bauerfeind I, Fehm T, Fleige B, Hausschild M, Helms G, Lebeau A, Liedtke C, von Minckwitz G, Nekljudova V, Schmatloch S, Schrenk P, Staebler A, Untch M. Sentinel-lymph-node biopsy in patients with breast cancer before and after neoadjuvant chemotherapy (SENTINA): a prospective, multicentre cohort study. Lancet Oncol. 2013 Jun;14(7):609-18. doi: 10.1016/S1470-2045(13)70166-9. Epub 2013 May 15. PMID 23683750
- [Result] Boileau JF, Poirier B, Basik M, Holloway CM, Gaboury L, Sideris L, Meterissian S, Arnaout A, Brackstone M, McCready DR, Karp SE, Trop I, Lisbona A, Wright FC, Younan RJ, Provencher L, Patocskai E, Omeroglu A, Robidoux A. Sentinel node biopsy after neoadjuvant chemotherapy in biopsy-proven node-positive breast cancer: the SN FNAC study. J Clin Oncol. 2015 Jan 20;33(3):258-64. doi: 10.1200/JCO.2014.55.7827. Epub 2014 Dec 1. PMID 25452445